CLINICAL TRIAL: NCT06431932
Title: Pharmacokinetics, Safety, and Efficacy of Fisetin - A Phase I and Pilot Phase IIa Study
Brief Title: Pilot Trial of Fisetin in Healthy Volunteers and Older Patients With Multimorbidity
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ove Andersen (Other)
Collaborators: University of Southern Denmark (Other); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, Head of Research, Clinical Professor, Principal Investigator, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fisetin; 2023-506284-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Multimorbidity; Healthy
Keywords: Senolytic; Pharmacokinetics; Chronic inflammation
MeSH Terms: interventions — fisetin

STUDY DESIGN:
Intervention Model Description: The trial consists of:
  * a single-arm open-label study, in which healthy volunteers (n=20) will receive fisetin corresponding to 20 mg/kg/day for two consecutive days.
  * a 2-arm triple-blind randomized placebo-controlled study, in which older patients with multimorbidity (n=40) will receive either:
    * 20 mg/kg/day fisetin for two consecutive days, or
    * placebo for two consecutive days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Single-arm open-label study in healthy volunteers (Experimental): Healthy volunteers will receive fisetin.
  Interventions: Drug: Fisetin
- RCT - Treatment group (Experimental): Older patients with multimorbidity will receive fisetin.
  Interventions: Drug: Fisetin
- RCT - Placebo group (Placebo Comparator): Older patients with multimorbidity will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — Subjects will receive fisetin corresponding to 20 mg/kg/day for two consecutive days.
  Arms: RCT - Treatment group; Single-arm open-label study in healthy volunteers
Drug: Placebo — Subjects will receive a corresponding number of placebo capsules for two consecutive days.
  Arms: RCT - Placebo group

SUMMARY:
The accumulation of senescent cells with age is a central mechanism that contributes to the development of chronic diseases, primarily by driving systemic chronic inflammation. Senolytic compounds such as fisetin can selectively target senescent cells for elimination and reduce multiple age-related pathologies in animal models.

We will conduct a clinical trial in healthy volunteers and older patients with multiple chronic diseases. The participants will receive fisetin or placebo for two days, after which they will be examined at regular intervals for up to three months. We will investigate how fisetin is absorbed and metabolized by the body, and whether fisetin is safe. We will also identify methods to best measure the effect of fisetin on chronic inflammation, senescent cells, and general health.

DETAILED DESCRIPTION:
The goal of this pilot trial is to conduct a controlled clinical study to gather data on the pharmacokinetic profile of fisetin and its metabolites and on the safety and tolerability of fisetin in healthy volunteers as well as in older medical patients. Furthermore, we aim to identify potential outcome measures and perform sample size calculations for these outcomes, with the intent to conduct a larger scale effect study, at later date, given the result from this pilot study suggests that this would be feasible and safe.

The trial consists of:

* a single-arm open-label study, in which healthy volunteers (n=20) will receive fisetin corresponding to 20 mg/kg/day for two consecutive days.
* a 2-arm triple-blind randomized placebo-controlled study, in which older medical patients (n=40) will receive either:

  * 20 mg/kg/day fisetin for two consecutive days, or
  * placebo for two consecutive days.

Each of the studies (open-label study and randomized placebo-controlled study) consists of three sub-studies:

* Sub-study I aims to investigate the pharmacokinetic properties of fisetin and its main metabolites following oral administration at a dose of 20 mg/kg/day in healthy volunteers and in older medical patients.
* Sub-study II aims to assess the safety and tolerability of oral treatment with fisetin at a dose of 20 mg/kg/day fisetin for two consecutive days in healthy volunteers and in older medical patients.
* Sub-study III aims to gather representative measurements to assess the utility of inflammation, SASP, senescence, senolysis, and aging biomarkers, as well as measures of frailty, clinical parameters, physical and cognitive function, and quality of life as potential outcomes in future clinical trials; additionally, to perform sample size calculations for future trials based on these data.

ELIGIBILITY:
Healthy volunteers:

Inclusion Criteria:

* Aged 20-35 years
* suPAR levels <3.5 ng/mL (± 15% corresponding to assay variation)
* Able to cooperate cognitively
* Able to read and understand Danish
* Women of childbearing potential must use effective contraception

Exclusion Criteria:

* Body weight >100 kg
* Inability to swallow pills
* Pregnant and/or lactating
* Known hypersensitivity or allergy to fisetin or excipients in the placebo capsules
* Presence of any condition that the investigator believes would put the subject at risk or would preclude the participant from successfully completing all aspects of the trial
* Presence of known chronic diagnosis
* Active acute illness
* Prescribed medication, except contraceptives
* Previous cancer diagnosis or treatment
* Use of senolytic and other "anti-aging" supplements

Older patients with multimorbidity:

Inclusion Criteria:

At screening #1 during hospital admission:

* Acutely hospitalized medical patient
* Age ≥65 years
* suPAR >5 ng/mL (± 15% corresponding to assay variation)
* Multimorbidity (≥2 chronic diagnoses)
* Able to cooperate cognitively
* Able to read and understand Danish

At screening #2 28 days after hospital discharge:

* suPAR >5 ng/mL (± 15% corresponding to assay variation)

Exclusion Criteria:

At screening #1 during hospital admission:

* Body weight >100 kg
* Inability to swallow pills
* Known human immunodeficiency virus infection, active hepatitis B or C infection, invasive fungal infection
* Uncontrolled (as per clinical judgment) pleural/pericardial effusions or ascites
* New/active invasive cancer except non-melanoma skin cancers
* Active cancer treatment or disseminated cancer
* Known condition associated with major immunodeficiency
* Known hypersensitivity or allergy to fisetin or excipients in the placebo capsules
* Use of senolytic and other "anti-aging" supplements

At screening #2 28 days after hospital discharge:

* Body weight >100 kg
* CRP >30 mg/L (± 15% corresponding to assay variation)
* Inability to swallow pills
* Presence of any condition, or abnormal routine biochemistry test, that the investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial
* Unstable (as per clinical judgment) major disorders, e.g., cardiovascular, renal, endocrine, immunological, hepatic disorder, or cancer
* Estimated glomerular filtration rate (eGFR) <15 ml/min/1.73 m2 or as per clinical judgment (e.g., risk of acute kidney injury)
* Human immunodeficiency virus infection, known active hepatitis B or C infection, invasive fungal infection
* Uncontrolled (as per clinical judgment) pleural/pericardial effusions or ascites
* New/active invasive cancer except non-melanoma skin cancers
* Active cancer treatment or disseminated cancer
* Known condition associated with major immunodeficiency
* Known hypersensitivity or allergy to fisetin or excipients in the placebo capsules
* Subjects taking strong inhibitors or inducers of CYP3A4 or as per clinical judgment
* Subjects taking specified substrates with a narrow therapeutic range for CYP3A4 or as per clinical judgment
* Subjects taking specified inhibitors, inducers, or substrates of CYP2D6, CYP2C9, or CYP2C8, or as per clinical judgment
* Subjects regularly using drug classes or specific medications or as per clinical judgment
* Use of senolytic and other "anti-aging" supplements

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Population-based pharmacokinetic model for fisetin and metabolites | 24 hours
  To develop a population-based pharmacokinetic (popPK) model for fisetin and its main metabolites in healthy volunteers and older patients, covariates such as body weight, body composition, age, and CYP inducers/inhibitors will be tested for influence on interindividual variability.
Adverse events | Day 1 to 3
  Number of participants to experience adverse events
suPAR | Day 1 to 29
  The change in plasma levels of suPAR and a sample size calculation based on these data.

SECONDARY OUTCOMES:
Population-based PKPD model for fisetin | 24 hours
  Changes in any of the measured biomarkers and the relationship between the pharmacokinetics and pharmacodynamics of fisetin will be investigated using population PKPD modeling.
Renal excretion of fisetin and its main metabolites | 24 hours
  Urinary levels of fisetin and its main metabolites
Symptoms and adverse events | Day 1 to 3
  Number of participants to experience symptoms and clinically significant changes in vital signs (i.e., blood pressure, pulse).
SASP factors and inflammation markers | Healthy volunteers: day 1, 2, 29. Older patients: day 1, 2, 8, 15, 29, 57, 84.
  The change in plasma levels of SASP factors and inflammation markers (e.g., cytokines, chemokines, proteases, growth factors).
Senescence | Healthy volunteers: day 1, 29. Older patients: day 1, 8, 15, 29, 84.
  The change in expression levels of senescence markers (e.g., p16INK4a, p21CIP1/WAF1, SA-B-gal) in immune cells and tissue biopsies (skin and adipose tissue).
Senolysis | Healthy volunteers: day 1, 2, 29. Older patients: day 1, 2, 8, 15, 29, 84.
  The change in expression levels of senolysis markers (e.g., leukotriene B4, dihomo-15d-PGJ2 (oxylipin or 1a,1b-dihomo-15-deoxy-D12,14-prostaglandin J2), and 15-Deoxy-delta 12, 14-prostaglandin J2).
Aging markers | Healthy volunteers: day 1, 2, 29. Older patients: day 1, 2, 8, 15, 29, 57, 84.
  The change in plasma levels of aging markers (e.g., α-klotho, fibroblast growth factor 21).
Clinical markers | Healthy volunteers: day 1, 2, 29. Older patients: day 1, 2, 8, 15, 29, 57, 84.
  The change in levels of routine biochemistry markers (e.g., alanine aminotransferase, albumin, alkaline phosphatase, bilirubin, blood urea nitrogen, coagulation factors II, VII and X and International Normalized Ratio, CRP, creatinine, hemoglobin, lactate dehydrogenase, mean corpuscular hemoglobin concentration, mean corpuscular volume, neutrophils, potassium, sodium, thrombocytes, white blood cell count, cholesterol (total, low-density lipoproteins, high-density lipoproteins), triglycerides, and hemoglobin A1c).
Frailty Index OutRef | Healthy volunteers: day 1, 29. Older patients: day 1, 2, 8, 15, 29, 57, 84.
  The change in frailty status calculated as Frailty Index OutREF (FI-OutRef).
Frailty Index | Healthy volunteers: day 1, 29. Older patients: day 1, 2, 8, 15, 29, 57, 84.
  The change in frailty status calculated using a modified version of Fried frailty criteria.
Physical function | Healthy volunteers: day 1, 29. Older patients: day 1, 29, 84.
  The change in physical function (e.g., gait speed, hand grip strength, chair stand test, balance).
Cognitive function (Montreal Cogntive Assessment) | Healthy volunteers: day 1, 29. Older patients: day 1, 29, 84.
  The change in cognitive function assessed using the MoCA score (0-30 with higher scores representing better cognitive function).
Cognitive function (Digit Symbol Substitution Test) | Healthy volunteers: day 1, 29. Older patients: day 1, 29, 84.
  The change in cognitive function assessed using the Digit Symbol Substitution Test (number of correct symbols).
Quality of life | Healthy volunteers: day 1, 29. Older patients: day 1, 29, 84.
  The change in quality of life assessed using the EuroQol-5D-5L (index value and VAS scale 0-100; with higher scores representing better quality of life).
Self-rated health | Healthy volunteers: day 1, 29. Older patients: day 1, 29, 84.
  The change in self-rated health (score 1-5; 1:"excellent", 2:"very good", 3:"good", 4:"fair", or 5:"bad").

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Tavenier, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Line Jee Hartmann Rasmussen, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Morten B Houlind, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Ove Andersen, Principal Investigator — Copenhagen University Hospital, Amager and Hvidovre; Jan O Nehlin, Study Chair — Copenhagen University Hospital, Amager and Hvidovre

IPD SHARING:
Plan to Share IPD: No
Only aggregated data can be available for other researchers due to Danish Data Protection Law.